CLINICAL TRIAL: NCT04239989
Title: A Phase I Study to Assess Safety of Selective JAK 1 Inhibitor, Itacitinib, in Patients With Bronchiolitis Obliterans Syndrome (BOS) After Allogeneic Hematopoietic Cell Transplant (HCT)
Brief Title: Itacitinib for the Treatment of Bronchiolitis Obliterans Syndrome After Donor Hematopoietic Cell Transplant
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: <75% participation
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0489; NCI-2019-08252 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0489 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-12-30; First posted 2020-01-27 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Bronchiolitis Obliterans
MeSH Terms: conditions — Bronchiolitis Obliterans | interventions — itacitinib; INCB039110

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (itacitinib) (Experimental): Patents receive itacitinib PO QD for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Itacitinib; Drug: Itacitinib Adipate

INTERVENTIONS:
Drug: Itacitinib — Given PO
  Other Names: INCB 039110; INCB-039110; INCB039110
Drug: Itacitinib Adipate — Given PO
  Other Names: INCB-039110 Adipate; INCB039110 Adipate

SUMMARY:
This phase I trial studies how well itacitinib works for the treatment of bronchiolitis obliterans syndrome after donor hematopoietic cell transplant. Itacitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the safety of itacitinib in patients with bronchiolitis obliterans syndrome (BOS) after allogeneic hematopoietic cell transplantation (HCT).

SECONDARY OBJECTIVES:

I. To assess treatment failure at 3 months and 6 months.

II. To assess change in symptom-based lung score at 3 months and 6 months.

III. To assess change in the St. George Respiratory Questionnaire and Study Short Form 36 at 3 months and 6 months.

IV. To assess change in the Lee chronic graft versus host disease (GVHD) symptom scale at 3 months and 6 months post-treatment.

V. To assess change in 6-minute walk test at 3 months and 6 months.

VI. To assess failure-free survival at 6 months.

VII. To assess non-relapse mortality at 6 months.

VIII. To assess overall survival at 6 months.

OUTLINE:

Patents receive itacitinib orally (PO) once daily (QD) for up to 1 year in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion criteria:

1. BOS diagnosed within the past 6 months of enrollment, defined by 2015 National Institutes of Health (NIH) Consensus Criteria 126
2. Age 18-75 years
3. Undergone allogeneic SCT
4. ANC >1,000/µL, hemoglobin > 8 gm/dL (untransfused) and platelet count >25,000/ µL (untransfused)
5. Karnofsky performance score >60
6. The ability to understand and sign a written informed consent form
7. Contraception for women and men of child bearing potential. Permitted methods should be at least 99% effective in preventing pregnancy.
8. Male patients must be willing to refrain from donating sperm during their participation in the study and for at least 3 months after completing the study.

Exclusion Criteria:

1. Prior treatment with any other JAK inhibitor (including Ruxolitinib) for BOS or any other indication within the past 6 months of enrolment.
2. Patients on mechanical ventilation or resting by pulse oximetry O2 saturation <88%
3. FEV1 <40% predicted
4. Relapsed primary malignancy for which SCT was performed
5. History of progressive multifocal leuko-encephalopathy (PML)
6. Active uncontrolled bacterial, fungal, parasitic, or viral infection
7. Known human immunodeficiency virus (HIV) infection or active hepatitis B or C infections.
8. History of tuberculosis anytime after SCT
9. Severe renal dysfunction defined by serum creatinine > 2 mg/dL, creatinine clearance <60 mL/minute or dialysis dependence
10. Serum transaminases > 5 × upper limit of normal
11. inability to perform PFT reliably
12. Positive Beta HCG test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization.
13. Lactating/nursing women
14. Life expectancy < 6 months
15. Other severe organ dysfunction unrelated to underlying GVHD. For example, uncontrolled or significant cardiac disease, including any of the following: recent myocardial infarction (within last 6 months from randomization); New York Heart Association Class III or IV congestive heart failure; unstable angina (within last 6 months prior to randomization); clinically significant (symptomatic) cardiac arrhythmias (e.g., sustained ventricular; tachycardia, and clinically significant second or third degree AV block without a pacemaker); uncontrolled hypertension. Or any other concurrent severe and/or uncontrolled medical conditions which, in the opinion of the investigator, could compromise participation in the study, pose a significant risk to the subject, or interfere with study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Monitoring the Dose Limiting Toxicities (DLT) of administering Itacitinib | Up to 6 months
  Number of participants who develop DLT's after the administration of the study drug

SECONDARY OUTCOMES:
Treatment failure | At 3 and 6 months
  Defined as a decrease in the absolute value of % forced expiratory volume in 1 second (FEV1) by 10% or more.
Changes in National Institutes of Health (NIH) symptom-based lung score | At 3 and 6 months
  Improvement in NIH symptom-based lung score; Score 0 (no symptoms), Score 1 (shortness of breath with stairs), Score 2 (shortness of breath on flat ground), and Score 3 (shortness of breath at rest or requiring oxygen
Change in well-established patient reported outcomes used in chronic graft versus host disease (GVHD) studies | Baseline and at 3 and 6 months
  Will include the St. George's Respiratory Questionnaire (SGRQ Regression models will include time, and different covariance structures will be included, including unstructured and autoregressive integrated moving average (ARIMA). The analysis will be adjusted for potential confounding variables. Participants will answer a St. George's Respiratory Questionnaire. (Very Poor, Poor, Fair, Good, Very Good)?
Change in well-established patient reported outcomes used in chronic graft versus host disease (GVHD) studies | Baseline up to 6 months
  Will include the Lee chronic GVHD symptom scale Lee symptom scale. Regression models will include time, and different covariance structures will be included, including unstructured and autoregressive integrated moving average (ARIMA). The analysis will be adjusted for potential confounding variables. The Lee Chronic GVHD Symptom Scale is a 30 item instrument with 7 subscales (skin, eyes, mouth, lung, nutrition, energy and psych) containing 2-7 items. Response options range from 0-4 (0-Not at all, 1-Slightly, 2-Moderately, 3-Quite a bit, 4-Extremely).
Change in well-established patient reported outcomes used in chronic graft versus host disease (GVHD) studies | Baseline and at 3 and 6 months
  Will include the study Short Form 36 (SF-36), NIH lung symptom score and SF-36 due to the longitudinal nature of the observations. Regression models will include time, and different covariance structures will be included, including unstructured and autoregressive integrated moving average (ARIMA). The analysis will be adjusted for potential confounding variables.
Change in 6-minute walk test | Baseline and at 3 and 6 months
Failure-free survival | At 6 months
  Will be assessed and monitored
Non-relapse mortality | At 6 months
  Defined as the absence of need for additional line treatment, non-relapse mortality and recurrent malignancy.
Overall survival | At 6 months
  Will be assessed and monitored

CONTACTS AND LOCATIONS:
Overall Officials: Amin Alousi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/89/NCT04239989/ICF_000.pdf